CLINICAL TRIAL: NCT03235674
Title: A Feasible High Intensity Interval Exercise Training Intervention in Phase II Cardiac Rehabilitation
Brief Title: Stair Climbing Outcomes in Cardiac Rehabilitation Exercise
Acronym: SCORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SCORE
Record Dates: First submitted 2017-06-09; First posted 2017-08-01 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2019-08

CONDITIONS: Endothelial Dysfunction
Keywords: Cardiac rehabilitation; interval exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity stair climbing exercise (Experimental): 3 x 60 seconds of stair climbing, at a vigorous pace as described by rating of perceived exertion, separated by 60 seconds of rest. Subjects will complete supervised sessions 3 times/week for 2 weeks, and then continue unsupervised for the following 10 weeks.
  Interventions: Other: High-intensity stair climbing exercise
- standard cardiac rehabilitation exercise (No Intervention): Subjects will complete the traditional cardiac rehabilitation program, combination of aerobic and resistance exercise 2 times/week for 2 weeks, and then continue unsupervised for the following 10 weeks.

INTERVENTIONS:
Other: High-intensity stair climbing exercise — High intensity stair climbing exercise at a vigorous pace as measured by rating of perceived exertion.
  Arms: High-intensity stair climbing exercise

SUMMARY:
This study will evaluate the effect of brief, intermittent stair climbing exercise on key cardiovascular and metabolic markers of health in individuals completing a cardiac rehabilitation program. Participants of this study will be placed into one of two exercise groups: one group will perform the standard exercise protocol currently being used by the Cardiac Health and Rehabilitation Centre at Hamilton General Hospital and the second group will perform a variation of interval exercise training, high intensity interval stair climbing.

DETAILED DESCRIPTION:
Cardiac rehabilitation (CR) is a recognized health service for the secondary prevention of CVD, unfortunately, CR is vastly underutilized, due to low referral rates and patient-related factors such as time commitment, travelling distance or user fees. After 2 weeks of CR exercise prescription, ~80% of patients opt to exercise independently rather than join a structured rehabilitation program in the community, suggesting that alternatives for current centre-based CR should focus on at-home programming with the intention of enhancing adherence and maintaining the lifestyle benefits long-term. The implementation of high-intensity interval exercise in CR programming has proven to be time-effective, enjoyable, safe, and capable of inducing similar if not superior cardiorespiratory responses, when compared to traditional, continuous CR programs. Recently, the benefits of interval stair climbing exercise in sedentary women were established, in that completing 3, 60 second bouts of high intensity stair climbing, 3 days/week for 6 weeks improved cardiorespiratory fitness, and represents a model of low-volume high-intensity interval training which is tolerable, effective and easily accessible for sedentary adults.

ELIGIBILITY:
Inclusion Criteria:

* Men and (post-menopausal) women
* Registered to participate in the Cardiac Health and Rehabilitation Centre (CHRC) at the Hamilton Health Sciences General Division
* History of previous myocardial infarction, coronary artery bypass graft, and/or percutaneous coronary intervention
* Non-smoker (within 3-months)
* Local resident, with transportation to the CHRC at the Hamilton Health Sciences General Division.
* Ability to understand written and verbal instructions and provide written informed consent.
* Stable medical therapy.

Exclusion Criteria:

* Non-cardiac surgical procedure within two months
* Positive exercise stress test (i.e. typical symptoms of chest discomfort and ECG changes or positive nuclear scan)
* Myocardial infarction within two months; coronary artery bypass graft surgery within two months; percutaneous coronary intervention within one month
* Baseline work capacity < 25 W
* NYHA class II-IV symptoms of heart failure
* Documented significant valve stenosis
* Symptomatic peripheral arterial disease that limits exercise capacity
* Uncontrolled supraventricular or ventricular dysrhythmia
* Unstable angina
* Uncontrolled hypertension (blood pressure >160/90 mmHg)
* Documented chronic obstructive pulmonary disease (FEV1 <60% and/or FVC <60%)
* Any musculoskeletal abnormality that would limit exercise participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
brachial endothelial function as measured by flow-mediated dilation (FMD) | Change from baseline FMD at 12 weeks
  This technique involves the placement of a blood pressure cuff around the forearm distal to the olecranon process (elbow). The cuff is inflated above systolic blood pressure to ~200 mmHg (in order to attain cessation of arm blood flow) and is held at this pressure for a period of five minutes. Continual measures of brachial artery diameter and blood flow velocity will be obtained using Doppler ultrasound. A 10 MHz probe will be placed on the upper arm (below the biceps) and moved around until the best signal is found. Images of brachial artery diameter and blood flow velocity will be taken at rest (before cuff inflation), prior to cuff deflation (end of five minute ischemic period), and following cuff deflation for two minutes.

SECONDARY OUTCOMES:
cardiorespiratory fitness | Change from baseline stress test at 12 weeks
  Maximal aerobic capacity will be determined using a medically monitored exercise stress test.
skeletal muscle capillary content | change from baseline capillary content at 12 weeks
  Muscle capillaries will be detected in frozen cross-sections of muscle biopsies based on positive staining with fluorescent lectin Ulex europaeus, and quantified relative to muscle fibre number (capillary:fibre ratio).
cardiac diastolic function | change from baseline left ventricular values at 12 weeks
  The heart must be imaged at both the base (top) and apex (bottom) of the left ventricle. Images will be taken in the parasternal short axis view with the participant lying in the left lateral decubitus position to allow the expansion of the rib cage and proper orientation of the heart within the chest cavity. Doppler ultrasound (5MHz sector probe) will be applied to the upper-middle section of the chest for the best images. Basal images will be taken at the tips of the mitral valves, while apical images will be taken at the most distal aspect of the left ventricle, with the LV cavity representing ~50% of the left ventricle wall thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen J MacDonald, PhD, Principal Investigator — McMaster University
Locations (1):
- Cardiac Health and Rehabilitation Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allison MK, Baglole JH, Martin BJ, Macinnis MJ, Gurd BJ, Gibala MJ. Brief Intense Stair Climbing Improves Cardiorespiratory Fitness. Med Sci Sports Exerc. 2017 Feb;49(2):298-307. doi: 10.1249/MSS.0000000000001188. PMID 28009784
- [Background] Aamot IL, Karlsen T, Dalen H, Stoylen A. Long-term Exercise Adherence After High-intensity Interval Training in Cardiac Rehabilitation: A Randomized Study. Physiother Res Int. 2016 Mar;21(1):54-64. doi: 10.1002/pri.1619. Epub 2015 Feb 16. PMID 25689059
- [Derived] Valentino SE, Dunford EC, Dubberley J, Lonn EM, Gibala MJ, Phillips SM, MacDonald MJ. Cardiovascular responses to high-intensity stair climbing in individuals with coronary artery disease. Physiol Rep. 2022 May;10(10):e15308. doi: 10.14814/phy2.15308. PMID 35591811
- [Derived] Dunford EC, Valentino SE, Dubberley J, Oikawa SY, McGlory C, Lonn E, Jung ME, Gibala MJ, Phillips SM, MacDonald MJ. Brief Vigorous Stair Climbing Effectively Improves Cardiorespiratory Fitness in Patients With Coronary Artery Disease: A Randomized Trial. Front Sports Act Living. 2021 Feb 16;3:630912. doi: 10.3389/fspor.2021.630912. eCollection 2021. PMID 33665614
- [Derived] Lim C, Dunford EC, Valentino SE, Oikawa SY, McGlory C, Baker SK, Macdonald MJ, Phillips SM. Both Traditional and Stair Climbing-based HIIT Cardiac Rehabilitation Induce Beneficial Muscle Adaptations. Med Sci Sports Exerc. 2021 Jun 1;53(6):1114-1124. doi: 10.1249/MSS.0000000000002573. PMID 33394901